CLINICAL TRIAL: NCT02346266
Title: SMART (School-aged Children Making Healthy Choices And Recognizing sTroke): A Pilot Trial of a Stroke Awareness Program
Brief Title: SMART (School-aged Children Making Healthy Choices And Recognizing sTroke)
Acronym: SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Los Amigos Research and Education Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 176
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Stroke
Keywords: Stroke; Stroke Prevention; Children; Education
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART (Active Comparator): The intervention group of school-aged children will receive education on the F.A.S.T. (Face, Arm, Speech and Time) acronym, additional signs and symptoms of stroke and the need for immediate activation of Emergency Medical Services (EMS) by calling 911.
  Interventions: Other: SMART Education
- Usual Care (No Intervention): This group will not receive stroke education.

INTERVENTIONS:
Other: SMART Education
  Arms: SMART

SUMMARY:
A stroke awareness program for school-aged children to learn the signs/symptoms of stroke, teach their parents and make healthy life-style choices.

DETAILED DESCRIPTION:
1. To educate school-aged children, grades 9th through 12th on the F.A.S.T. (Face, Arm, Speech and Time) acronym, additional signs and symptoms of stroke and the need for immediate activation of Emergency Medical Services (EMS) by calling 911.
2. To improve adults' stroke literacy through educating their children in grades 9th through 12th.

ELIGIBILITY:
Inclusion Criteria:

* High-school student

Exclusion Criteria:

* Not a high-school student

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 480 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Child Improved Stroke Literacy | 3 weeks
  A school-based stroke literacy program targeting children in grades 9th through 12th will be successful in improving stroke literacy.

SECONDARY OUTCOMES:
Adult Improved Stroke Literacy | 3 weeks
  If school-aged children, grades 9th through 12th are taught the F.A.S.T. acronym, additional signs and symptoms of stroke and the immediate activation of EMS by calling 911, they will improve the stroke literacy of their parents.